CLINICAL TRIAL: NCT03152344
Title: Evaluation of a Simple Clinical Test to Detect the Risk of Falling in Patients With Chronic Obstructive Pulmonary Disease and Research for Predictive Factors of Fall Risk.
Brief Title: Evaluation of a Simple Clinical Test to Detect the Risk of Falling in Patients With BPCO and Research for Predictive Factors of Fall Risk.
Acronym: Equil-BPCO
Status: Completed | Type: Observational
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: Centre de Recherche en Nutrition Humaine d'Auvergne (Other Government)
Responsible Party: Sponsor
Other Study IDs: CHU-332; 2016-A01188-43 (Other: 2016-A01188-43)
Record Dates: First submitted 2017-05-11; First posted 2017-05-15 (Actual); Last update posted 2019-08-13 (Actual); Status verified 2019-08

CONDITIONS: COPD Diagnosed
Keywords: Fall; Balance control; Screening test; Oxygen; Skeletal muscle mass

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- COPD patients without chronic respiratory failure: We will recruit COPD patients in stable condition (free of exacerbation of the disease for a month), 40 without chronic respiratory failure and 40 with home oxygen therapy.
  The patients will be proposed to perform the following tests and to fill in questionnaires
  Interventions: Procedure: Timed Up and Go
- COPD patients with home oxygen therapy: We will recruit COPD patients in stable condition (free of exacerbation of the disease for a month), 40 without chronic respiratory failure and 40 with home oxygen therapy.
  The patients will be proposed to perform the following tests and to fill in questionnaires
  Interventions: Procedure: Timed Up and Go

INTERVENTIONS:
Procedure: Timed Up and Go — It's a functional test evaluating the time to rise from a chair, walk 3 meters, turn around, walk back to the chair and sit down (abnormal cut-off value >12 seconds).

SUMMARY:
The risk of falling in increased in patients with Chronic Obstructive Pulmonary Disease. To date, a screening test (the Berg Balance scale, BBS) is used to evaluate this risk but it spends 20 to 30 minutes to complete.

The aim of our study is to evaluate the sensitivity of a more straightforward test (Timed Up and Go, TUG)) to assess the fall risk. The TUG is routinely used in elderly to screen for frailty.

DETAILED DESCRIPTION:
We will recruit COPD patients in stable condition (free of exacerbation of the disease for a month), 40 without chronic respiratory failure and 40 with home oxygen therapy.

The patients will be proposed to perform the following tests and to fill in questionnaires:

- Questionnaires: Elderly Falls Screening Test to quantify the falls in the last year, Hospital Anxiety and Depression Scale, Activities-specific Balance Confidence scale.

Tests:

* Berg Balance Scale measuring balance in 14 different functional tasks (abnormal cut-off value <56)
* Timed Up and Go evaluating the time to rise from a chair, walk 3 meters, turn around, walk back to the chair and sit down (abnormal cut-off value >12 seconds).
* 6 minute walk test evaluating endurance to submaximal exercise.
* Isokinetic maximal force of the quadriceps at 60°/s
* Balance control: posturography consisting in measuring variations when standing on a force platform.
* Body composition assessment through Dual Xray Absorptiometry (DXA), to measure body muscle mass and more specifically appendicular muscle mass index as a criteria of sarcopenia, and bone mineral density.
* Blood analysis: a blood sample will be withdrawn to measure calcium, phosphorus, vitamin D, albumin transthyretin, cell count, C reactive protein.

Analysis of the results:

We will calculate the sensitivity of the TUG test (abnormal test) to detect fall risk as assessed by an abnormal BBS score.

Moreover, in fallers, we will search for predictive factors. More specifically, we will look for the role of a decreased quadriceps force, a reduced muscle mass, a poor tolerance of exercise, the presence of hypoxia (severity of the disease).

Perspectives:

When validated as a screening test for the risk of falling in COPD patients, the TUG test could be used routinely by physiotherapists as a more simple and faster test and will enable to prevent falls through initiation of a balance control training program.

ELIGIBILITY:
Inclusion Criteria:

* COPD confirmed by pulmonary function tests
* Long term oxygen therapy since at least 3 months in the LOT+ subgroup

Exclusion Criteria:

* Exacerbation of COPD necessitating an hospitalization or an oral corticosteroid treatment, in the last 4 weeks
* Pulmonary rehabilitation in the last 3 months
* Any neurological disease affecting balance control.
* Inability to perform a walk test

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We will recruit COPD patients in stable condition (free of exacerbation of the disease for a month), 40 without chronic respiratory failure and 40 with home oxygen therapy.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2017-01-02 (Actual); Primary Completion 2017-10-27 (Actual); Study Completion 2017-10-27 (Actual)

PRIMARY OUTCOMES:
Comparison of the Timed Up and Go test and the Berg Balance scale | at day 1
  Comparison of the consistency of abnormal value of the Timed Up and Go test and the Berg Balance scale

SECONDARY OUTCOMES:
Sensitivity of the TUG test and the BBS | at day 1
  to detect fall as assessed by the Elderly Falls Screening Test.
Difference in BBS score | at day 1
  between COPD patients without and with chronic respiratory failure (LOT+/- subgroups).
Identify predictive factors of fall risk | at day 1
  walk distance, quadriceps force, muscle mass, balance control.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Clermont-Ferrand, Clermont-Ferrand, Auvergne, France